CLINICAL TRIAL: NCT04995172
Title: Mobile-CT-Assisted Bronchoscopy
Brief Title: Feasibility of Mobile-CT-Assisted Bronchoscopy for the Diagnosis of Lung Lesion
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0760; NCI-2021-01331 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0760 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-07-28; First posted 2021-08-06 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Lung Neoplasm
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (CT-assisted bronchoscopy, chart review): Patients undergo RP-EBUS bronchoscopy per standard of care. If the study staff cannot reach the target lesion or is unable to determine a diagnosis, patients undergo bronchoscopy using mobile CT imaging. Patients' medical records are also reviewed for up to 6 months.
  Interventions: Procedure: Computed Tomography; Other: Electronic Health Record Review; Procedure: Endobronchial Ultrasound Bronchoscopy

INTERVENTIONS:
Procedure: Computed Tomography — Undergo mobile CT-assisted bronchoscopy
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Electronic Health Record Review — Patients' medical records are reviewed
Procedure: Endobronchial Ultrasound Bronchoscopy — Undergo radial probe EBUS
  Other Names: EBUS; Endobronchial Ultrasound

SUMMARY:
This study investigates whether using a mobile-CT-assisted bronchoscopy (M-CAB) during a bronchoscopy procedure will better enable the study staff to reach the lung tumor, perform a biopsy, and obtain a diagnosis. One method that doctors use for diagnosing lung tumors is bronchoscopy guided by an X-ray machine (called fluoroscope). Though much better guidance could be provided with a CT scanner when compared to the fluoroscope, the standard CT equipment is very large, fixed in a radiology room, and difficult to use with bronchoscopy. Mobile CT imaging systems may more easily and effectively perform the same tasks of the standard CT imaging in the bronchoscopy room, offering better guidance than the standard fluoroscope.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE

I. To determine the added value of mobile-CT)-assisted bronchoscopy (M-CAB) for the diagnosis of peripheral lung nodules defined as the proportion of patients in whom bronchoscopy with radial-probe endobronchial ultrasound (RP-EBUS) and 2-D Fluoroscopy is non-diagnostic (lesion is not reached or rapid-onsite cytology is non-diagnostic) and diagnosis is obtained after utilizing mobile-CT assistance.

SECONDARY OBJECTIVES:

I. Describe the navigational yield of bronchoscopy with RP-EBUS/2-dimensional (2-D) fluoroscopy for peripheral nodules.

II. Describe the diagnostic yield of bronchoscopy with RP-EBUS/2-D fluoroscopy for peripheral nodules.

III. Describe the mobile-CT (M-CT) added navigational yield. IV. Describe the sensitivity for malignancy of bronchoscopy with RP-EBUS/2-D fluoroscopy and its increase (if any) provided by mobile-CT assistance.

V. Describe anatomical and procedural characteristics that can influence navigational and diagnostic yield (tumor location, tumor characteristics -solid, semisolid-, air-bronchus sign, biopsy tool, relationship between biopsy tool/tumor).

VI. Describe procedure duration. VII. Describe time required to obtain mobile CT scans VIII. Describe fluoroscopy time and estimate radiation dose to the patient. IX. Describe procedural complications.

OUTLINE:

Patients undergo RP-EBUS bronchoscopy per standard of care. If the study staff cannot reach the target lesion or is unable to determine a diagnosis, patients undergo bronchoscopy using mobile CT imaging. Patients' medical records are also reviewed for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years of age or older undergoing bronchoscopy for diagnosis of a peripheral lung lesion from 1 to 3.5 cm in diameter located in the outer 2/3 of the lung fields

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients who cannot tolerate raising both arms above their head (position for obtaining mobile-CT images)
* Patients with any contraindication for general anesthesia (e.g., severe and active coronary artery disease, chronic obstructive pulmonary disease (COPD) with forced expiratory volume in 1 second (FEV1) < 1 liter, uncontrolled hypertension, increased intracranial pressure, history of intolerance to general anesthesia)
* Dementia or other severe cognitive impairment causing inability to understand or consent to the procedure and study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with a peripheral lung lesion who are scheduled to undergo a bronchoscopy
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
The added value of mobile-computed tomography (CT)-assisted bronchoscopy (M-CAB) | Up to 6 months
  Defined as the proportion of patients in whom bronchoscopy with thin or ultrathin scope, radial-probe endobronchial ultrasound (RP-EBUS) and 2-dimensional (2-D) fluoroscopy is non-diagnostic (lesion is not reached or rapid-onsite cytology is non-diagnostic) and diagnosis is obtained after utilizing mobile-CT assistance. Descriptive statistics (mean standard deviation [SD] or median interquartile range [IQR], frequency [%]) will be used to summarize patient characteristics.

SECONDARY OUTCOMES:
Navigational yield of thin/ultrathin scope/RP-EBUS/2-D fluoroscopy for peripheral nodules | Up to 6 months
  Navigational yield for standard of care (SOC) will be estimated along with 95% confidence intervals (CIs).
Diagnostic yield of thin/ultrathin scope/RP-EBUS/2-D fluoroscopy for peripheral nodules | Up to 6 months
  Diagnostic yield of SOC and diagnostic yield of SOC + M-CT along with their 95% CIs will be estimated.
Mobile-CT (M-CT) added navigational yield | Up to 6 months
  M-CT added diagnostic yield in a subgroup with non-diagnostic subjects by SOC will be estimated along with its 95% CI. M-CT added diagnostic yield in a subgroup with non-diagnostic subjects by SOC will be estimated along with its 95% CI. Two-sided exact binomial test will be used to test if diagnostic yield of SOC + M-CT is significantly different from 0.2 in the subgroup.
Sensitivity for malignancy of thin/ultrathin scope/RP-EBUS/2-D fluoroscopy and its increase (if any) provided by mobile-CT assistance | Up to 6 months
  Sensitivity for malignancy of SOC and sensitivity for malignancy of SOC + M-CT will be estimated, considering final pathology as the gold standard test.
Anatomical and procedural characteristics that can influence navigational and diagnostic yield | Up to 6 months
  Anatomic and procedural characteristics that are associated with navigational and diagnostic yield will be evaluated by multivariate logistic regression models. A p-value of less than 0.05 will indicate a statistical significance.
Procedure duration | Up to 6 months
  Will be summarized by mean (standard deviation [SD]) or median (interquartile range [IQR]).
Time required to obtain mobile CT scans | Up to 6 months
  Will be summarized by mean (SD) or median (IQR).
Fluoroscopy time | Up to 6 months
  Will be summarized by mean (SD) or median (IQR).
Radiation dose to the patient | Up to 6 months
  Will be summarized by mean (SD) or median (IQR).
Procedural complications | Up to 6 months
  Complications will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto F Casal, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org